CLINICAL TRIAL: NCT06457919
Title: A Phase 1b/2 Study Evaluating the Activity of Tinengotinib (TT-00420) in Combination With Androgen Receptor Signaling Inhibitors (ARSIs) in Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: A Study of Tinengotinib (TT-00420) in Combination With Standard Treatments in People With Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: TransThera Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-103
Record Dates: First submitted 2024-06-05; First posted 2024-06-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
Keywords: Tinengotinib (TT-00420); Androgen Receptor Signaling Inhibitors (ARSIs); TIP Study: Tinengotinib In Prostate Cancer; Prostate Cancer Clinical Trials Consortium, LLC (PCCTC); 24-103
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone; enzalutamide

STUDY DESIGN:
Intervention Model Description: In the Phase 1b portion of the study, participants will be enrolled sequentially in cohorts of 3 for each studied combination. The recommended Phase II dose (RP2D) of each combination will be estimated separately based on the de-escalation rules.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tinengotinib with abiraterone acetate/prednisone (Experimental): Tinengotinib will be administered daily for 28-day cycles. A flat dose of 10 mg PO once daily will be administered unless dose de-escalation is required in Phase 1b. Participants will receive tinengotinib with abiraterone acetate 1000 mg PO QD in combination with prednisone 5 mg PO once or twice daily (QD or BID)
  Interventions: Drug: Tinengotinib; Drug: abiraterone acetate with prednisone
- Tinengotinib with enzalutamide (Experimental): Tinengotinib will be administered daily for 28-day cycles. A flat dose of 10 mg PO once daily will be administered unless dose de-escalation is required in Phse 1b. Participants will receive Tinengotinib in combination with enzalutamide 160 mg PO QD.
  Interventions: Drug: Tinengotinib; Drug: Enzalutamide

INTERVENTIONS:
Drug: Tinengotinib — Tinengotinib will be administered daily for 28-day cycles. A flat dose of 10 mg PO once daily.
  Other Names: TT-00420
Drug: abiraterone acetate with prednisone — Abiraterone acetate 1000 mg PO QD in combination with prednisone 5 mg PO once or twice daily (QD or BID)
  Arms: Tinengotinib with abiraterone acetate/prednisone
Drug: Enzalutamide — Enzalutamide 160 mg PO QD
  Arms: Tinengotinib with enzalutamide

SUMMARY:
The purpose of this study is to find out whether tinengotinib in combination with abiraterone acetate and prednisone or enzalutamide is a safe treatment that causes few or mild side effects in people with metastatic castration-resistant prostate cancer (mCRPC).

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥ 18 years old, with signed informed consent
* Histologically confirmed carcinoma of the prostate (neuroendocrine differentiation is allowed, but pure small cell carcinoma is not permitted)
* Metastatic disease documented by at least 2 bone lesions on whole body radionuclide bone scan, or soft tissue disease documented by computed tomography (CT) scan/magnetic resonance imaging (MRI). Note: Metastatic disease seen only on PET imaging does not qualify.
* Current ongoing therapy and observed tolerance with full standard dose of abiraterone acetate (1000 mg QD) or enzalutamide (160 mg QD) at the time of study entry. Enzalutamide or abiraterone acetate must have been started at least 90 days before screening assessments. An interruption of dosing of a maximum of 30 days is permitted prior to resuming the agent. Please note: Patients who are on a reduced dose or are intolerant of abiraterone acetate or enzalutamide at screening will not be eligible for study participation.
* Progressive disease on enzalutamide or abiraterone acetate documented by PCWG3 criteria for study entry. Progressive disease is defined as at least one of the following:

  1. PSA progression defined as a minimum of 2 rising PSA levels with a minimum of a 1-week interval between each determination, reaching a minimum PSA value of 1.0 ng/mL.
  2. Nodal or visceral progression as defined by PCWG3-modified RECIST 1.1
  3. Appearance of 2 or more new lesions on a bone scan
* At least one of the following at study entry:

  1. RECIST 1.1 measurable disease at baseline; i.e., soft tissue tumor lesions or pathologically enlarged lymph nodes that can be accurately measured in at least one dimension OR
  2. a PSA of 2.0 ng/mL or above
* Participants must be medically or surgically castrated with ongoing androgen deprivation therapy (ADT) for ≥90 days or have documented history of bilateral orchiectomy.
* ECOG 0 - 2
* Adequate organ function confirmed at screening, as evidenced by:

  * Absolute neutrophil count ≥ 1.5 × 10^9 /L
  * Hemoglobin ≥ 9 g/dL
  * Platelets ≥ 75 × 10^9 /L
  * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 2.5 × upper limit of normal (ULN) or ≤ 5.0 × ULN if liver metastases are present
  * Total bilirubin ≤ 1.5 × ULN; or < 2.5 × ULN if Gilbert syndrome or disease involving liver
  * Creatinine clearance >30 mL/min (Cockcroft-Gault formula)
  * Adequate blood coagulation function as evidence by an international normalized ratio (INR) ≤ 1.5 unless participant is on anticoagulants
* Tumor biopsy during screening is required if safe and feasible. If archival tissue is available from a previous biopsy performed within 90 days of screening assessments, a repeat screening biopsy is not required even if safe and feasible. If neither option is possible, archival tissue from any timepoint should be requested, if available.

Exclusion Criteria:

* The presence of any of the following criteria excludes a patient from participating in the study:
* Pure small cell carcinoma
* Previous exposure to multi-TKI therapies.
* Uncontrolled hypertension (persistent systolic blood pressure ≥ 140 mm Hg and/or diastolic blood pressure ≥ 90 mm Hg) or known coronary artery disease with angina. Patients with known hypertension must be on antihypertensive medication with BPs generally <140/90 to be eligible.
* History of congestive heart failure of Class II-IV New York Heart Association criteria, or serious cardiac arrhythmia requiring treatment (except atrial fibrillation, paroxysmal supraventricular tachycardia), history of myocardial infarction within 6 months of study entry, or prolongation of QTc interval to >480 msec using Fridericia formula (QTcF) at screening (except for participants with pacemakers, where there is no QTc cutoff).
* Any prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessments.
* Symptomatic and/or untreated CNS metastases.
* Pre-existing duodenal stent or any gastrointestinal disorder or defect which would interfere with absorption of study medication, as determined by the Investigator.
* Persistent requirement for corticosteroids at equivalent of >10 mg QD prednisone within 14 days before study treatment start.
* Other anticancer therapies within 3 weeks of study treatment start, or within 5 half-lives of study treatment start for non-cytotoxic oral agents, whichever is shorter; with the exception of androgen deprivation therapy, enzalutamide, or abiraterone acetate which should be continued through study treatment.
* Palliative radiation within 2 weeks of study treatment start.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 50 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
RP2D | From the start of study treatment through the DLT window (28 days)
  Evaluate DLT occurrence to confirm safety and RP2D
Objective Response Rate (ORR) | up to 6months
  by local investigator's assessment per PCWG3-modified RECIST v1.1 in participants with baseline measurable disease OR rate of PSA decline of ≥ 50% from baseline in patients with a baseline PSA of 2.0 ng/mL or above

SECONDARY OUTCOMES:
Rate of Radiographic Response (phase II) | From start of study treatment until 6 months post study treatment start
  Rate of radiographic response by local investigator's assessment per PCWG3-modified RECIST v1.1 in participants with baseline measurable disease

CONTACTS AND LOCATIONS:
Overall Officials: Wassim Abida, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (11):
- United States (11):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Columbia University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York
  - Duke University, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm